CLINICAL TRIAL: NCT04423055
Title: Nexplanon Use in Women Primarily Choosing a Combined Oral Contraceptive: a Multicenter Trial
Brief Title: Nexplanon Use in Women Primarily Choosing a Combined Oral Contraceptive
Acronym: NextOC2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); University of Colorado, Denver (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1571368
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2023-06

CONDITIONS: Contraception
Keywords: Contraceptive implant; Nexplanon; Combined oral contraceptive
MeSH Terms: interventions — etonogestrel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- COC users or new starts (Experimental): Subjects will have an etonogestrel contraceptive implant placed at enrollment. Women using COC as method of contraception for at least 1 month will be considered COC users. Women using COC for less than 1 month will be considered new starts.
  Interventions: Drug: Etonogestrel contraceptive implant

INTERVENTIONS:
Drug: Etonogestrel contraceptive implant — Place etonogestrel contraceptive implant.
  Other Names: Nexplanon

SUMMARY:
Women currently using or starting a combined oral contraceptive (COC) will be offered study enrollment. Study subjects will have a Nexplanon placed and followed for approximately 12 months to evaluate if they continue the implant, the COC, or both, and to assess bleeding patterns and adverse events.

DETAILED DESCRIPTION:
This study will be conducted at three sites across the United States: University of California, Davis, University of Colorado and University of Pennsylvania. Investigators will recruit women currently using COCs or intending to initiate COCs for pregnancy prevention. Each site will recruit approximately 40 women for a total of 120 subjects.

Visit 1:

Informed consent will be obtained. As part of informed consent, subjects will be educated that there is little data available on the adverse effects of combined COC and ENG implant use. The consent form will include a standardized description of the side effects and bleeding profile of COCs and the implant. Subjects will also need to review the package label information for Nexplanon and sign the FDA-required Nexplanon consent. After obtaining informed consent, subjects will be screened for entry criteria. Medical history will be obtained. A urine pregnancy test will be performed. Eligible subjects will have a Nexplanon contraceptive implant placed. A diary will be dispensed for the subject to document daily bleeding, COC use and adverse events.

Follow-up:

Follow up contact will be at approximately 4, 12, 26 and 39 weeks with the exit visit scheduled at 52 weeks.

At each follow up contact, the diary will be reviewed. Adverse events will be determined by inquiry and diary review. The subject will inform the study staff if she is using her COC and if she wants to continue use of her COC and ENG implant. The ENG implant will be removed upon request at any time during the study.

Study participation will be complete after the 52 week (~ 12 month) exit visit.

No blood draws will occur during this study.

A diary will be used but no surveys will be used.

Data to be collected by study staff include demographics, past medical and gynecologic history, prior and current contraceptive use.

Because women are being enrolled who are already currently using COCs or who plan to start COCs, the COC is not a study drug. The study intervention (study drug) is the contraceptive implant. The systemic hormone exposure with a contraceptive implant is minimal relative to a COC. The investigators do not expect any increase in side effects by adding a contraceptive implant to COC users. Of note, the primary risk with COC use is related to the estrogen which can increase the risk of venous thromboembolic disease. The implant has no estrogen. All products being used in the study are FDA-approved for contraception.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years and older currently using COCs or who have a COC prescription and are intending to initiate COCs for contraception

Exclusion Criteria:

* Women who have contraindications to using a COC or a contraceptive implant (Category 3 or 4 in the CDC Medical Eligibility Criteria [MEC])
* Because the CDC MEC are continuously revised, the most updated criteria will be used (http://www.cdc.gov/mmwr/preview/mmwrhtml/rr5904a3.htm)
* Women who are currently participating in a clinical trial or have participated within the past 30 days.
* Less than 2 weeks from the end of a pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants Evaluating ENG Implant as Acceptable | 52 weeks
  Evaluate the acceptability (continuation of the implant throughout the study) of concomitant etonogestrel (ENG) implant use in women choosing a combined oral contraceptive (COC) for contraception

SECONDARY OUTCOMES:
Number of Participants Evaluating ENG as Tolerable: Tolerability | 52 weeks
  Evaluate the tolerability (side effects) of concomitant etonogestrel (ENG) implant use in women choosing a combined oral contraceptive (COC) for contraception
Number of Participants Continuing COC | 52 weeks
  Continuation of COC over 52 weeks of evaluation regardless of whether or not the implant was still present at 52 weeks
Bleeding Patterns | 52 weeks
  Bleeding patterns while using a COC concomitantly with ENG implant
Post-study Method Plan | 52 weeks
  Plan to continue the COC and/or implant after the study based on interview at last visit

CONTACTS AND LOCATIONS:
Overall Officials: Melissa C Matulich, MD MAS, Principal Investigator — University of California, Davis
Locations (3):
- United States (3):
  - University of California, Davis, Sacramento, California
  - University of Colorado, Denver, Colorado
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No